CLINICAL TRIAL: NCT06782672
Title: Investigation of Objective Cognitive Effort in Neuropsychological Evaluation of Psychotic Disorders
Acronym: INVESTIGECCO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: fondation john bost (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHLMPL23_0456
Record Dates: First submitted 2024-12-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Psychotic Disorders; Cognitive Impairment; Motivation
Keywords: memory; effort; cardiovascular reactivity
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psychotic disorders: The target population is people with a psychotic disorder (diagnosed as schizophrenia or schizoaffective disorder) according to DSM 5 criteria, aged between 18 and 60.
  The people with psychotic disorders recruited for this study are currently being cared for at the adult psychiatry department of Montpellier University Hospital.
  Participants will have a single visit with memory tests and data recording (cardiovascular, performance, perceptions), followed by a psychological assessment using questionnaires and a semi-structured interview.
  Interventions: Other: Cardiovascular measurements; Other: Experimental memory task; Other: Questionnaire and semi-structured psychological interview
- non clinical, control: The non-clinical population should be similar to the psychotic disorders population in terms of age, level of education and gender.
  Participants will have a single visit with memory tests and data recording (cardiovascular, performance, perceptions), followed by a psychological assessment using questionnaires and a semi-structured interview.
  Interventions: Other: Cardiovascular measurements; Other: Experimental memory task; Other: Questionnaire and semi-structured psychological interview

INTERVENTIONS:
Other: Cardiovascular measurements — Measurement of pre-ejection period is the period between the onset of electrical excitation of the left ventricle and the opening of the aortic valve and heart rate will be continuous.
  These data will be collected using a cardiograph measuring the ECG signal and impedance cardiography (ICG). The system's four electrodes are positioned on the middle axillary line at the end of the sternum and at the base of the neck.
  Blood pressure measurements (PAS and PAD) will be taken from a cuff placed on the brachial artery of the non-dominant arm.
  cardiovascular values will be measured continuously:
  * Each participant rested while watching a documentary for 8 minutes.
  * During two 5-minute memory tasks of different difficulty levels (easy and difficult), separated by a 5-minute break.
  The averages of the last 5 minutes during the resting period will constitute the resting values, and the averages of the 5 minutes of each difficulty level will constitute the values during cognitive effort.
Other: Experimental memory task — First, a quiet period with the viewing of a documentary film (8min).
  Then, participants will perform two 5-minute memory tasks of different difficulty levels (memorizing 3 letters corresponds to the easy level vs. 7 letters to the difficult level), separated by a 5-minute break. The order of difficulty will be counterbalanced.
  At the end of each difficulty level, self-report measures assessed by the following questions will be collected:
  * "How much effort did you exert during the task?";
  * How difficult did you find the task?
  * How motivated were you to perform the task? Responses will be in Likert scale format, ranging from 1 ("no effort at all", "very easy", "not at all motivated", respectively) to 7 ("a lot of effort", "very difficult", "very motivated", respectively).
Other: Questionnaire and semi-structured psychological interview — psychopathological measures collected using questionnaires:
  * Beck Depression Inventory (BDI-II): mood
  * State-Trait Anxiety Inventory (Form Y) (STAY-Y): anxiety
  * Multidimensional Fatigue Inventory, 20-item version (MFI-20=): fatigue
  * General Self-Efficacy Scale (GSES): defeatist beliefs
  * Clinical Assessment Interview for Negative Symptoms (CAINS) : psychotic symptoms for the psychotic disorders group

SUMMARY:
Psychotic disorders are characterised by a heterogeneity of symptoms, including cognitive disorders, which predict functional outcome. To date, the evaluation of cognitive functions essentially measures performance. Cognitive effort and the influence of psychological factors are rarely considered.

Based on the principle of energy conservation, the Motivational Intensity Theory (MIT) allows to test cognitive effort independently of performance, by measuring cardiovascular reactivity, as well as controlling for psychological factors (e.g., mood, fatigue, anxiety).

The main aim of this study is to investigate in a memory task the interaction between cognitive effort, performance and psychological factors in individuals with psychotic disorders compared to a non-clinical group, based on the predictions of the MIT.

This study will provide insights into the nature of cognitive impairment in psychotic disorders: primary or secondary to motivational (effort) or psychological (mood, fatigue, anxiety) difficulties.

DETAILED DESCRIPTION:
The study will be proposed to patients with psychotic disorders (n=50) and non clinical participants (n = 50) aged 18 to 60.

This is a non-interventional, randomized, prospective experimental study with mixed design: 2 groups (psychotic disorders vs. non-clinical) with 2 repeated measures of difficulty (easy vs. difficult).

The study comprises a single visit with memory tests recording cardiovascular, and performance data, as well as participants' perceptions of the task (effort invested, difficulty, motivation to perform the task), followed by a psychological assessment using questionnaires and a semi-structured interview.

The study of these different measures (cardiovascular, performance, perception) will enable us to refine the understanding of cognitive deficits in psychotic disorders, taking psychopathological variables into account. will provide better direction for the care of this population: cognitive remediation for primary cognitive disorders vs. cognitive and behavioral therapies for cognitive disorders secondary to psychopathological variables (mood, fatigue, defeatist beliefs, motivational deficits).

ELIGIBILITY:
Inclusion Criteria in both groups

- Age ≥ 18 years and ≤60 years

Inclusion criteria for the psychotic disorders group:

- Patients with a diagnosis within the schizophrenia spectrum and other psychotic disorders according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5; APA, 2015).

Inclusion criterion for the non-clinical group:

- Absence of any psychiatric disorder.

non-inclusion criteria in both groups

* Neurological disorder or history of head trauma;
* Cardiovascular disease or treatment for hypertension;
* Substance abuse or dependence disorder;
* Individuals who cannot understand or speak French;
* Non-affiliation with a social security system;
* Individuals participating in another study that includes an ongoing exclusion period;
* Individuals who have not provided written informed consent to participate in the study;
* Pregnant or breastfeeding women;
* Absence of written consent from the legal guardian for patients under guardianship;
* Absence of notification to the curator for patients under curatorship.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Non-clinical group: Absence of any psychiatric disorder, community sample
  Psychotic disorders group : Patients with a diagnosis within the schizophrenia spectrum and other psychotic disorders according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5; APA, 2015), selected from the adult psychiatry department, inpatient or outpatient hospitalisation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-27 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Interaction effect of group x difficulty on cardiovascular reactivity (Pre-Ejection Period - PEP) | 18 minutes
  The difference score between the pre-ejection period (PEP) during the task (easy and difficult) and the PEP at rest (i.e., baseline), expressed in ms.

SECONDARY OUTCOMES:
Investigation of systolic blood pressure in both groups and difficulties | 18 minutes
  expressed in mmHg
Investigation of diastolic blood pressure in both groups and difficulties | 18 minutes
  expressed in mmHg
Investigation of heart rate pressure in both groups and difficulties | 18 minutes
  expressed in beats/minutes
Comparison of correct performance | 10 minutes
  The percentage of correct responses between the two groups and in both levels of difficulty
Comparison of errors | 10 minutes
  The rate of errors between the two groups and in both levels of difficulty
Comparison of self-reported effort in both groups and both difficulties | 1 minute
  Self-reported effort will assess through the following question:
  - "How much effort did you exert during the task?" Response will be on a Likert scale ranging from 1 ('Not at all effort') to 7 ('A lot of effort').
Comparison of self-reported difficulty in both groups and both difficulties | 1 minute
  Self-reported difficulty will assess through the following question:
  "How difficult did you find the task?" Response will be on a Likert scale ranging from 1 ('Very easy') to 7 ('Very difficult').
Comparison of self-reported motivation in both groups and both difficulties | 1 minute
  Self-reported motivation will assess through the following question:
  "How motivated were you to complete the task?" Response will be on a Likert scale ranging from 1 ('Not at all motivated') to 7 ('Very motivated').
Influence of depressed mood on effort | 5 minutes
  Beck Depression Inventory (BDI-II, Beck et al., 1996, internal consistency α = .92). This self-administered questionnaire consists of 21 items, each scored from 0 to 3. The total score ranges from 0 to 63.
  The higher the score, the more severe the depression.
Influence of anxiety on effort | 5 minutes
  State-Trait Anxiety Inventory (Form Y) (STAY-Y, Spielberger et al., 1983, Bruchon-Schweitzer & Paulhan, 1993 for French validation, internal consistency α = .91). The STAY-Y assesses two scales momentary anxiety and trait anxiety, each comprising 20 items. Scores range from 1 ("Not at all for the momentary anxiety scale, "Almost never" for the trait anxiety scale) to 4 ("A lot", "Almost always", respectively). The higher the score, the more severe the anxiety.
Influence of fatigue on effort | 3 minutes
  Multidimensional Fatigue Inventory, 20-item version (IMF-20, Smets et al., 1995, Gentille et al., 2003 for French validation, internal consistency α > .70). This scale comprises 20 items ranging from 1 ("Strongly disagree") to 5 ("Strongly agree").The total score is between 4 and 20, the higher the score, the greater the fatigue felt.The MFI has 5 subscales: general fatigue, mental fatigue, reduced motivation, physical fatigue, reduced activities.
Influence of defeatist beliefs on effort | 3 minutes
  General Self-Efficacy Scale (GSES, Schwarzer & Jerusalem, 1995, Dumont et al., 2000, for French validation, internal consistency α > .76).This scale measures feelings of self-efficacy . This scale measures feelings of self-efficacy (the opposite of defeatist beliefs). It comprises 10 items, scored on a Likert scale ranging from 1 ("Not at all true") to 4 ("Totally true"). The higher the score, the higher the sense of self-efficacy, and the lower the person's self-defeating beliefs.
Influence of negatives symptomes on effort in schizophrenia group | 30 minutes
  Clinical Assessment Interview for Negative Symptoms (CAINS, Kring et al., 2013; Laraki et al., 2022 for French validation, internal consistency α = 0.87). This is a semi-structured interview assessing the negative symptoms of schizophrenia.
  This interview is composed of 13 items ranging from 0 (absence/no deficit) to 5 (severe deficit). The interview includes two subscales: motivation and pleasure (MAP, 9 items) and expressivity (EXP, 4 items).

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Décombe, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided